CLINICAL TRIAL: NCT02065791
Title: A Randomized, Double-blind, Event-driven, Placebo-controlled, Multicenter Study of the Effects of Canagliflozin on Renal and Cardiovascular Outcomes in Subjects With Type 2 Diabetes Mellitus and Diabetic Nephropathy
Brief Title: Evaluation of the Effects of Canagliflozin on Renal and Cardiovascular Outcomes in Participants With Diabetic Nephropathy
Acronym: CREDENCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: The George Institute for Global Health, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR103517; 2013-004494-28 (EudraCT Number); 28431754DNE3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2014-02-17; First posted 2014-02-19 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2; Diabetic Nephropathy
Keywords: Diabetes Mellitus, Type 2; Diabetic Nephropathies; Canagliflozin; JNJ-28431754; End-Stage Kidney Disease; Chronic Kidney Disease; Macroalbuminuria
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Canagliflozin 100 mg (Experimental): Each participant will receive 100 mg of canagliflozin once daily
  Interventions: Drug: Canagliflozin
- Placebo (Placebo Comparator): Each participant will receive matching placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — One 100 mg over-encapsulated tablet orally once daily
  Arms: Canagliflozin 100 mg
Drug: Placebo — One matching placebo capsule orally (by mouth) once daily
  Arms: Placebo

SUMMARY:
The goal of this study is to assess whether canagliflozin has a renal and vascular protective effect in reducing the progression of renal impairment relative to placebo in participants with type 2 diabetes mellitus (T2DM), Stage 2 or 3 chronic kidney disease (CKD) and macroalbuminuria, who are receiving standard of care including a maximum tolerated labeled daily dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB).

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the identity of the assigned treatment), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect), parallel-group, multicenter study of the effects of canagliflozin on renal and cardiovascular outcomes in participants with type 2 diabetes mellitus (T2DM) and diabetic nephropathy, who are receiving standard of care including a maximum tolerated daily dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB).

The study will consist of a pretreatment phase (several weeks), and a double-blind treatment phase (up to approximately 66 months). During the pretreatment phase all participants will also receive diet/exercise counseling for lipid and blood pressure management as well as counseling on renal and cardiovascular (CV) risk factor medication. A post-treatment follow-up contact or visit will take place approximately 30 days after the last dose of study drug or the completion of the study. The total duration of the study is estimated to be about 5 to 5.5 years. Approximately 4,200 participants will be randomized in a 1:1 ratio to canagliflozin or matching placebo. Participants randomized to canagliflozin will receive a dose of 100 mg once daily. The overall safety and tolerability of canagliflozin will be evaluated by collecting information on adverse events, laboratory tests, vital signs (pulse, blood pressure), physical examination, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus with a hemoglobin A1c (HbA1c) greater than or equal to (>=) 6.5 percent (%) and less than or equal to (<=) 12.0%, with an estimated glomerular filtration rate (eGFR) of >= 30 milliliter (mL)/minute (min)/1.73meter (m)^2 and less than (<) 90 mL/min/1.73 m^2
* Participants need to be on a stable maximum tolerated labeled daily dose of an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin receptor blocker (ARB) for at least 4 weeks prior to randomization
* Must have a urine albumin to creatinine ratio (UACR) of greater than (>) 300 milligram (mg)/gram (g) and <= 5000 mg/g

Exclusion Criteria:

* History of diabetic ketoacidosis or type 1 diabetes mellitus
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Renal disease that required treatment with immunosuppressive therapy
* Known significant liver disease
* Current or history of New York Heart Association (NYHA) Class IV heart failure
* Blood potassium level >5.5 millimole (mmol)/liter (L) during Screening

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4401 (Actual)
Dates: Start 2014-02-17 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (575):
- United States (152):
  - Birmingham, Alabama
  - Montgomery, Alabama
  - Tempe, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Sherwood, Arkansas
  - Bakersfield, California
  - Chula Vista, California
  - Covina, California
  - Downey, California
  - Fountain Valley, California
  - Hawthorne, California
  - Inglewood, California
  - Laguna Hills, California
  - Lakewood, California
  - Long Beach, California
  - Los Angeles, California
  - Lynwood, California
  - Northridge, California
  - Oakland, California
  - Orange, California
  - Pasadena, California
  - Roseville, California
  - Sacramento, California
  - Salinas, California
  - San Diego, California
  - San Dimas, California
  - Stanford, California
  - Tustin, California
  - Whittier, California
  - Denver, Colorado
  - Golden, Colorado
  - Lakewood, Colorado
  - Washington, Colorado
  - Washington D.C., District of Columbia
  - Coral Springs, Florida
  - Doral, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Springs, Florida
  - North Miami Beach, Florida
  - Ocala, Florida
  - Port Charlotte, Florida
  - St. Petersburg, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Columbus, Georgia
  - Roswell, Georgia
  - Snellville, Georgia
  - Stockbridge, Georgia
  - Chicago, Illinois
  - Crystal Lake, Illinois
  - Gurnee, Illinois
  - Mount Prospect, Illinois
  - Winfield, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Merrillville, Indiana
  - Michigan City, Indiana
  - Muncie, Indiana
  - Council Bluffs, Iowa
  - Louisville, Kentucky
  - Paducah, Kentucky
  - Kenner, Louisiana
  - Rockport, Maine
  - Scarborough, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Beltsville, Maryland
  - Hyattsville, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Plymouth, Massachusetts
  - Springfield, Massachusetts
  - Worcester, Massachusetts
  - Flint, Michigan
  - Jackson, Mississippi
  - Chesterfield, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Fremont, Nebraska
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Reno, Nebraska
  - Las Vegas, Nevada
  - Eatontown, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Binghamton, New York
  - Buffalo, New York
  - Great Neck, New York
  - Lake Success, New York
  - New Hyde Park, New York
  - New York, New York
  - Ridgewood, New York
  - Riverhead, New York
  - Smithtown, New York
  - Springfield Gardens, New York
  - Asheville, North Carolina
  - Calabash, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - High Point, North Carolina
  - Morehead City, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Tabor City, North Carolina
  - Whiteville, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Maumee, Ohio
  - Roseburg, Oregon
  - Beaver, Pennsylvania
  - Bethlehem, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Anderson, South Carolina
  - Columbia, South Carolina
  - Lancaster, South Carolina
  - Murrells Inlet, South Carolina
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Arlington, Texas
  - Corpus Christi, Texas
  - Corsicana, Texas
  - Dallas, Texas
  - Edinburg, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Mesquite, Texas
  - San Antonio, Texas
  - Schertz, Texas
  - Sugar Land, Texas
  - Temple, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Burlington, Vermont
  - Bluefield, Virginia
  - Mechanicsville, Virginia
  - Norfolk, Virginia
  - Suffolk, Virginia
  - Spokane, Washington
  - Huntington, West Virginia
  - Milwaukee, Wisconsin
- Argentina (29):
  - Bahía Blanca
  - Buenos Aires
  - Ciudad Autonoma Buenos Aires
  - Corrientes
  - Córdoba
  - Godoy Cruz
  - Junín
  - La Plata
  - La Plata Lpl Lpl
  - Mar del Plata
  - Mendoza
  - Morón
  - Munro
  - Paraná
  - Quilmes
  - Ramos Mejía
  - Rosario
  - Salta
  - San Luis
  - San Martín
  - San Migeul de Tucuman
  - San Miguel de Tucumán
  - San Nicolás
  - Santa Fe
  - Sarandí
  - Tapiales
  - Temperley
  - Villa María
  - Zarate, Buenos Aires
- Australia (16):
  - Cairns
  - Concord
  - Darlinghurst
  - Elizabeth Vale
  - Fremantle
  - Gosford
  - Heidelberg
  - Keswick
  - Meadowbrook
  - Parkville
  - Reservoir
  - Richmond
  - St Albans
  - St Leonards
  - Sydney
  - Woolloongabba
- Brazil (22):
  - Aparecida de Goiânia
  - Belém
  - Belo Horizonte
  - Botucatu
  - Brasília
  - Campina Grande do Sul
  - Campinas
  - Canoas
  - Caxias do Sul
  - Curitiba
  - Fortaleza
  - Joinville
  - Juiz de Fora
  - Maringá
  - Passo Fundo
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
  - São José do Rio Preto
  - São José dos Campos
  - São Paulo
  - Tatuí
- Bulgaria (8):
  - Blagoevgrad
  - Byala
  - Golenci
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Sofia
  - Varna
- Canada (18):
  - Edmonton, Alberta
  - New Westminster, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Brampton, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - Oshawa, Ontario
  - Smiths Falls, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Weston, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Québec
  - Toronto
  - Vancouver
- Chile (3):
  - Concepción
  - Santiago
  - Temuco
- China (17):
  - Beijing
  - Changchun
  - Changde
  - Changsha
  - Chengdu
  - Chenzhou
  - Dalian
  - Foshan
  - Guangzhou
  - Huai'an
  - Nanchang
  - Nanjing
  - Shanghai
  - Shenyang
  - Ürümqi
  - Wuhan
  - Xi'an
- Colombia (9):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Cali
  - Floridablanca
  - Manizales
  - Medellín
  - Pasto
  - Pereira
- Czechia (13):
  - Choceň
  - České Budějovice
  - Český Krumlov
  - Havlíčkův Brod
  - Hradec Kralove-Vekose
  - Hradec nad Svitavou
  - Jindřichův Hradec
  - Olomouc
  - Prague
  - Slaný
  - Trutnov
  - Uherské Hradiště
  - Ústí nad Labem
- France (16):
  - Besançon
  - Brest
  - Colmar
  - Corbeil-Essonnes
  - Créteil
  - Grenoble
  - Lyon
  - Marseille
  - Metz
  - Nantes
  - Paris
  - Pierre-Bénit
  - Poitiers
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
- Germany (8):
  - Bad Kreuznach - Bosenheim
  - Cologne
  - Dietzenbach
  - Dresden
  - Essen
  - Hamburg
  - Hanover
  - Münster
- Guatemala City, Guatemala
- Hungary (18):
  - Baja
  - Balatonfüred
  - Budapest
  - Debrecen
  - Eger
  - Esztergom
  - Gödöllő
  - Gyula
  - Hu-4012 Debrecen N/a
  - Kaposvár
  - Kecskemét
  - Komárom
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szigetvár
  - Veszprém
  - Zalaegerszeg
- India (14):
  - Calicut
  - Chennai
  - Delhi
  - Hyderabad
  - Kozhikode
  - Lucknow
  - Ludhiyāna
  - Mangalore
  - Mumbai
  - Mysore
  - Secunderabad
  - Trivandrum
  - Vijayawada
  - Visakhapatnam
- Japan (26):
  - Ageo-shi
  - Chiyoda-ku
  - Fukuoka
  - Hamamatsu
  - Hamura-shi
  - Ina-shi
  - Izumisano
  - Kamakura-shi
  - Kanazawa
  - Kawanishi-shi
  - Koriyama-shi
  - Kuki-shi
  - Kyoto
  - Matsuyama
  - Midori
  - Minatoku
  - Nagoya
  - Osaka
  - Ota-shi
  - Saiki-shi
  - Sashima-gun
  - Shinjuku-ku
  - Toyama
  - Uwajima-shi
  - Yamanashi
  - Yokohama
- Lithuania (3):
  - Kaunas
  - Klaipėda
  - Šiauliai
- Malaysia (13):
  - Batu Caves
  - Ipoh
  - Johor Bahru
  - Kuala Lumpur
  - Kuantan
  - Malacca
  - Perai
  - Petaling Jaya
  - Seremban
  - Seri Manjung
  - Sungai Petani, Kedah
  - Tampin
  - Temerluh
- Mexico (22):
  - Aguascalientes
  - Celaya
  - Chihuahua City
  - Ciudad de Mexic
  - Cuautitlán Izcalli
  - Culiacán
  - Durango
  - El Salto
  - Guadalajara
  - León
  - Mexico City
  - Mérida
  - México
  - Monterrey
  - Morelia
  - Orizaba
  - Pachuca
  - Querétaro
  - San Luis Potosí City
  - Tlalnepantla
  - Veracruz
  - Zapopan
- New Zealand (8):
  - Auckland
  - Christchurch
  - Dunedin
  - Palmerston North
  - Rotorua
  - Takapuna Auckland
  - Tauranga
  - Wellington
- Philippines (13):
  - Cagayan de Oro
  - Cebu
  - Cebuu City
  - Davao City
  - Iloilo City
  - Lipa City
  - Marikina City
  - Pasay
  - Pasig
  - Quezon City
  - San Fernando City
  - Tagbilaran City
  - Taytay
- Poland (15):
  - Bydgoszcz
  - Chorzów
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Parczew
  - Poznan
  - Radom
  - Rzeszów
  - Torun
  - Warswa
  - Wroclaw
  - Zgierz
  - Żnin
- Puerto Rico (3):
  - Caguas
  - Ponce
  - San Juan
- Romania (9):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Deva
  - Iași
  - Oradea
  - Ploieşti
  - Târgu Mureş
  - Timișoara
- Russia (16):
  - Arkhangelsk
  - Barnaul
  - Ivanovo
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Sestroretsk, Saint-Petersburg
  - Tomsk
  - Ufa
  - Volgograd
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Niš
  - Zaječar
- Slovakia (11):
  - Bardejov
  - Bratislava
  - Košice
  - Ľubochňa
  - Nitra
  - Prievidza
  - Púchov
  - Rimavská Sobota
  - Svidník
  - Štúrovo
  - Žilina
- South Africa (9):
  - Cape Town
  - Durban
  - Isipingo Rail
  - Johannesburg
  - Krugersdorp
  - Port Elizabeth
  - Pretoria
  - Pretoria Gauteng
  - Soweto
- South Korea (5):
  - Busan
  - Daegu
  - Incheon
  - Seongnam
  - Seoul
- Spain (20):
  - A Coruña
  - Almería
  - Barcelona
  - Burela de Cabo
  - Ciudad Real
  - Getafe
  - Girona
  - Granada
  - La Roca del Vallès
  - Madrid
  - Majadahonda
  - Málaga
  - Palma de Mallorca
  - Pozuelo de Alarcón
  - Sagunto
  - Santander
  - Seville
  - Valencia
  - Vic
  - Viladecans
- Taiwan (4):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Taipei
- Ukraine (10):
  - Chernivtsi
  - Dnipropetrovsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Ternopil
  - Vinnitsya
  - Vinnytsia
  - Zaporizhzhia
- United Arab Emirates (3):
  - Ajman
  - Dubai
  - Sharjah city
- United Kingdom (38):
  - Aberdeen
  - Antrim
  - Barry
  - Birmingham
  - Blackburn
  - Bolton
  - Bournemouth
  - Bradford
  - Bristol
  - Burbage
  - Cardff
  - Cardiff
  - Carlshalton
  - Carmarthen
  - Chester
  - Darlington
  - Doncaster
  - Durham
  - Ely
  - Hampstead
  - Harlow
  - Huntingdon
  - Liskeard
  - London
  - Middlesbrough
  - Plymouth
  - Rhyl
  - Royal Leamington Spa
  - Rugby
  - Salford
  - Stoke-on-Trent
  - Swansea
  - Torpoint
  - Watford
  - Welwyn Garden City
  - Westcliff-on-Sea
  - Wokingham
  - Wolverhampton

REFERENCES:
- [Derived] Mottl A, Scott C, Green JB, Heerspink HJL, Mann JFE, McGill JB, Nangaku M, Rosenstock J, Rossing P, Li L, Li N, Vaduganathan M, Agarwal R; CONFIDENCE Trial Investigators. Baseline Kidney Function, Albuminuria, and Urine Albumin-Creatinine Ratio Reduction with Finerenone, Empagliflozin, or Both: Post Hoc Analyses of CONFIDENCE Trial. J Am Soc Nephrol. 2025 Nov 6. doi: 10.1681/ASN.0000000928. Online ahead of print. No abstract available. PMID 41196655
- [Derived] Bayes-Genis A, Cai A, Liu Y, Pandey A, Pop-Busui R, Hansen M, Januzzi JL. Impact of canagliflozin on heart stress and outcomes: Pooled insights from CREDENCE and CANVAS. Eur J Heart Fail. 2025 Dec;27(12):2887-2896. doi: 10.1002/ejhf.3786. Epub 2025 Jul 21. PMID 40689549
- [Derived] Oshima M, Buizen L, Jongs N, Levin A, Chertow GM, Wheeler DC, Heerspink HJL, Arnott C, Jardine MJ, Mahaffey KW, Pollock C, Herrington WG, Perkovic V, Neuen BL. Sodium-Glucose Cotransporter 2 Inhibition and Hospitalizations in Patients with CKD: A Meta-Analysis of Kidney Outcome Trials. Clin J Am Soc Nephrol. 2025 Jul 14;20(9):1206-1214. doi: 10.2215/CJN.0000000771. PMID 40658498
- [Derived] Jongs N, Gasparyan SB, Frison L, Schloemer P, Brinker M, Little DJ, Heerspink HJL. Use of eGFR Slope Thresholds as End Point Components in a Kidney Disease Progression Hierarchical Composite End Point. J Am Soc Nephrol. 2025 Dec 1;36(12):2421-2430. doi: 10.1681/ASN.0000000766. Epub 2025 Jun 17. PMID 40526444
- [Derived] Januzzi JLJ, Sattar N, Vaduganathan M, Magaret CA, Rhyne RF, Liu Y, Masson S, Butler J, Hansen MK. A validated multivariable machine learning model to predict cardio-kidney risk in diabetic kidney disease. Cardiovasc Diabetol. 2025 May 15;24(1):213. doi: 10.1186/s12933-025-02779-5. PMID 40375260
- [Derived] Doi Y, Hamano T, Yamaguchi O, Isaka Y. Canagliflozin may increase thromboembolic events in males with erythrocytosis but not in females. Blood Adv. 2025 Jul 8;9(13):3202-3212. doi: 10.1182/bloodadvances.2025016320. PMID 40239057
- [Derived] Nguyen TN, Yu J, Perkovic V, Jardine M, Mahaffey KW, Chow CK, Arnott C, Lindley RI. The Efficacy and Safety of Canagliflozin by Frailty Status in Participants of the CANVAS and CREDENCE Trials. J Am Geriatr Soc. 2025 Jun;73(6):1787-1796. doi: 10.1111/jgs.19444. Epub 2025 Mar 19. PMID 40105285
- [Derived] Chatur S, Vaduganathan M, Fletcher RA, Perkovic V, Heerspink H, Arnott C, Pollock C, Mahaffey KW, Neal B, Jardine M, Solomon SD, Neuen BL. Canagliflozin reduces oral loop diuretic intensification in patients with type 2 diabetes: A participant-level pooled analysis of the CANVAS and CREDENCE trials. Eur J Heart Fail. 2025 Jun;27(6):994-1002. doi: 10.1002/ejhf.3586. Epub 2025 Jan 23. PMID 39844714
- [Derived] Vaduganathan M, Cannon CP, Jardine MJ, Heerspink HJL, Arnott C, Neuen BL, Sarraju A, Gogate J, Seufert J, Neal B, Perkovic V, Mahaffey KW, Kosiborod MN. Effects of canagliflozin on total heart failure events across the kidney function spectrum: Participant-level pooled analysis from the CANVAS Program and CREDENCE trial. Eur J Heart Fail. 2024 Sep;26(9):1967-1975. doi: 10.1002/ejhf.3292. Epub 2024 Jun 26. PMID 38932575
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Januzzi JL Jr, Liu Y, Sattar N, Yavin Y, Pollock CA, Butler J, Jardine M, Heerspink HJL, Masson S, Breyer M, Hansen MK. Vascular endothelial growth factors and risk of cardio-renal events: Results from the CREDENCE trial. Am Heart J. 2024 May;271:38-47. doi: 10.1016/j.ahj.2024.02.016. Epub 2024 Feb 22. PMID 38401646
- [Derived] Sharma A, Razaghizad A, Joury A, Levin A, Bajaj HS, Mancini GBJ, Wong NC, Slee A, Ang FG, Rapattoni W, Neuen BL, Arnott C, Perkovic V, Mahaffey KW. Primary and Secondary Cardiovascular and Kidney Prevention With Canagliflozin: Insights From the CANVAS Program and CREDENCE Trial. J Am Heart Assoc. 2024 Feb 6;13(3):e031586. doi: 10.1161/JAHA.123.031586. Epub 2024 Jan 19. PMID 38240199
- [Derived] Mohebi R, Liu Y, Hansen MK, Yavin Y, Sattar N, Pollock CA, Butler J, Jardine M, Masson S, Heerspink HJL, Januzzi JL Jr. Associations of Angiopoietin 2 and Vascular Endothelial Growth Factor-A Concentrations with Clinical End Points. Clin J Am Soc Nephrol. 2024 Apr 1;19(4):429-437. doi: 10.2215/CJN.0000000000000389. Epub 2023 Dec 14. PMID 38099944
- [Derived] Fletcher RA, Jongs N, Chertow GM, McMurray JJV, Arnott C, Jardine MJ, Mahaffey KW, Perkovic V, Rockenschaub P, Rossing P, Correa-Rotter R, Toto RD, Vaduganathan M, Wheeler DC, Heerspink HJL, Neuen BL. Effect of SGLT2 Inhibitors on Discontinuation of Renin-angiotensin System Blockade: A Joint Analysis of the CREDENCE and DAPA-CKD Trials. J Am Soc Nephrol. 2023 Dec 1;34(12):1965-1975. doi: 10.1681/ASN.0000000000000248. Epub 2023 Oct 25. PMID 37876229
- [Derived] Heerspink HJL, Jongs N, Schloemer P, Little DJ, Brinker M, Tasto C, Karpefors M, Wheeler DC, Bakris G, Perkovic V, Nkulikiyinka R, Rossert J, Gasparyan SB. Development and Validation of a New Hierarchical Composite End Point for Clinical Trials of Kidney Disease Progression. J Am Soc Nephrol. 2023 Dec 1;34(12):2025-2038. doi: 10.1681/ASN.0000000000000243. Epub 2023 Oct 24. PMID 37872654
- [Derived] Yu J, Sweeting AN, Gianacas C, Houston L, Lee V, Fletcher RA, Perkovic V, Li Q, Neuen BL, Berwanger O, Heerspink HJL, de Zeeuw D, Arnott C. The effects of canagliflozin in type 2 diabetes in subgroups defined by population-specific body mass index: Insights from the CANVAS Program and CREDENCE trial. Diabetes Obes Metab. 2023 Dec;25(12):3724-3735. doi: 10.1111/dom.15267. Epub 2023 Sep 6. PMID 37671609
- [Derived] Januzzi JL, Mohebi R, Liu Y, Sattar N, Heerspink HJL, Tefera E, Vaduganathan M, Butler J, Yavin Y, Li J, Pollock CA, Perkovic V, Neal B, Hansen MK. Cardiorenal Biomarkers, Canagliflozin, and Outcomes in Diabetic Kidney Disease: The CREDENCE Trial. Circulation. 2023 Aug 22;148(8):651-660. doi: 10.1161/CIRCULATIONAHA.123.065251. Epub 2023 Aug 21. PMID 37603600
- [Derived] Mohebi R, Liu Y, Hansen MK, Yavin Y, Sattar N, Pollock CA, Butler J, Jardine M, Masson S, Heerspink HJL, Januzzi JL Jr. Insulin growth factor axis and cardio-renal risk in diabetic kidney disease: an analysis from the CREDENCE trial. Cardiovasc Diabetol. 2023 Jul 12;22(1):176. doi: 10.1186/s12933-023-01916-2. PMID 37438734
- [Derived] Fletcher RA, Arnott C, Rockenschaub P, Schutte AE, Carpenter L, Vaduganathan M, Agarwal R, Bakris G, Chang TI, Heerspink HJL, Jardine MJ, Mahaffey KW, Neal B, Pollock C, Jun M, Rodgers A, Perkovic V, Neuen BL. Canagliflozin, Blood Pressure Variability, and Risk of Cardiovascular, Kidney, and Mortality Outcomes: Pooled Individual Participant Data From the CANVAS and CREDENCE Trials. J Am Heart Assoc. 2023 Jul 4;12(13):e028516. doi: 10.1161/JAHA.122.028516. Epub 2023 Jun 22. PMID 37345834
- [Derived] Ferrannini G, Pollock C, Natali A, Yavin Y, Mahaffey KW, Ferrannini E. Extremes of both weight gain and weight loss are associated with increased incidence of heart failure and cardiovascular death: evidence from the CANVAS Program and CREDENCE. Cardiovasc Diabetol. 2023 Apr 29;22(1):100. doi: 10.1186/s12933-023-01832-5. PMID 37120538
- [Derived] van der Hoek S, Jongs N, Oshima M, Neuen BL, Stevens J, Perkovic V, Levin A, Mahaffey KW, Pollock C, Greene T, Wheeler DC, Jardine MJ, Heerspink HJL. Glycemic Control and Effects of Canagliflozin in Reducing Albuminuria and eGFR: A Post Hoc Analysis of the CREDENCE Trial. Clin J Am Soc Nephrol. 2023 Jun 1;18(6):748-758. doi: 10.2215/CJN.0000000000000161. Epub 2023 Mar 31. PMID 36999981
- [Derived] Yi TW, Smyth B, Di Tanna GL, Arnott C, Cardoza K, Kang A, Pollock C, Agarwal R, Bakris G, Charytan DM, de Zeeuw D, Heerspink HJL, Neal B, Wheeler DC, Cannon CP, Zhang H, Zinman B, Perkovic V, Levin A, Mahaffey KW, Jardine M; CREDENCE Trial Investigators. Kidney and Cardiovascular Effects of Canagliflozin According to Age and Sex: A Post Hoc Analysis of the CREDENCE Randomized Clinical Trial. Am J Kidney Dis. 2023 Jul;82(1):84-96.e1. doi: 10.1053/j.ajkd.2022.12.015. Epub 2023 Mar 7. PMID 36889425
- [Derived] Sarraju A, Bakris G, Cannon CP, Cherney D, Damaraju CV, Figtree GA, Gogate J, Greene T, Heerspink HJL, Januzzi JL Jr, Neal B, Jardine MJ, Blais J, Kosiborod M, Levin A, Lingvay I, Weir MR, Perkovic V, Mahaffey KW. Cardiovascular Effects of Canagliflozin in Relation to Renal Function and Albuminuria. J Am Coll Cardiol. 2022 Nov 1;80(18):1721-1731. doi: 10.1016/j.jacc.2022.08.772. PMID 36302584
- [Derived] Nunes JC, Yu J, Arnott C, Jardine MJ, Perkovic V, Mahaffey KW. Canagliflozin, mental health adverse events and diabetes: Exploratory analysis of the CREDENCE trial and CANVAS Program. Diabetes Obes Metab. 2022 Dec;24(12):2459-2464. doi: 10.1111/dom.14832. Epub 2022 Aug 19. No abstract available. PMID 35938182
- [Derived] Li JW, Arnott C, Heerspink HJL, MBiostat QL, Cannon CP, Wheeler DC, Charytan DM, Barraclough J, Figtree GA, Agarwal R, Bakris G, de Zeeuw D, Greene T, Levin A, Pollock C, Zhang H, Zinman B, Mahaffey KW, Perkovic V, Neal B, Jardine MJ. Effect of Canagliflozin on Total Cardiovascular Burden in Patients With Diabetes and Chronic Kidney Disease: A Post Hoc Analysis From the CREDENCE Trial. J Am Heart Assoc. 2022 Aug 16;11(16):e025045. doi: 10.1161/JAHA.121.025045. Epub 2022 Aug 5. PMID 35929472
- [Derived] Charytan DM, Yu J, Jardine MJ, Cannon CP, Agarwal R, Bakris G, Greene T, Levin A, Pollock C, Powe NR, Arnott C, Mahaffey KW; CREDENCE study investigators. Potential Effects of Elimination of the Black Race Coefficient in eGFR Calculations in the CREDENCE Trial. Clin J Am Soc Nephrol. 2022 Mar;17(3):361-373. doi: 10.2215/CJN.08980621. Epub 2022 Jan 21. PMID 35063969
- [Derived] Heerspink HJL, Oshima M, Zhang H, Li J, Agarwal R, Capuano G, Charytan DM, Craig J, de Zeeuw D, Di Tanna GL, Levin A, Neal B, Perkovic V, Wheeler DC, Yavin Y, Jardine MJ. Canagliflozin and Kidney-Related Adverse Events in Type 2 Diabetes and CKD: Findings From the Randomized CREDENCE Trial. Am J Kidney Dis. 2022 Feb;79(2):244-256.e1. doi: 10.1053/j.ajkd.2021.05.005. Epub 2021 May 23. PMID 34029680
- [Derived] Zhou Z, Jardine MJ, Li Q, Neuen BL, Cannon CP, de Zeeuw D, Edwards R, Levin A, Mahaffey KW, Perkovic V, Neal B, Lindley RI; CREDENCE Trial Investigators*. Effect of SGLT2 Inhibitors on Stroke and Atrial Fibrillation in Diabetic Kidney Disease: Results From the CREDENCE Trial and Meta-Analysis. Stroke. 2021 May;52(5):1545-1556. doi: 10.1161/STROKEAHA.120.031623. Epub 2021 Apr 20. PMID 33874750
- [Derived] Yu J, Li J, Leaver PJ, Arnott C, Huffman MD, Udell JA, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Matthews DR, Shaw W, Rosenthal N, Neal B, Figtree GA. Effects of canagliflozin on myocardial infarction: a post hoc analysis of the CANVAS programme and CREDENCE trial. Cardiovasc Res. 2022 Mar 16;118(4):1103-1114. doi: 10.1093/cvr/cvab128. PMID 33826709
- [Derived] Jardine M, Zhou Z, Lambers Heerspink HJ, Hockham C, Li Q, Agarwal R, Bakris GL, Cannon CP, Charytan DM, Greene T, Levin A, Li JW, Neuen BL, Neal B, Oh R, Oshima M, Pollock C, Wheeler DC, de Zeeuw D, Zhang H, Zinman B, Mahaffey KW, Perkovic V. Kidney, Cardiovascular, and Safety Outcomes of Canagliflozin according to Baseline Albuminuria: A CREDENCE Secondary Analysis. Clin J Am Soc Nephrol. 2021 Mar 8;16(3):384-395. doi: 10.2215/CJN.15260920. Epub 2021 Feb 22. PMID 33619120
- [Derived] Ye N, Jardine MJ, Oshima M, Hockham C, Heerspink HJL, Agarwal R, Bakris G, Schutte AE, Arnott C, Chang TI, Gorriz JL, Cannon CP, Charytan DM, de Zeeuw D, Levin A, Mahaffey KW, Neal B, Pollock C, Wheeler DC, Luca Di Tanna G, Cheng H, Perkovic V, Neuen BL. Blood Pressure Effects of Canagliflozin and Clinical Outcomes in Type 2 Diabetes and Chronic Kidney Disease: Insights From the CREDENCE Trial. Circulation. 2021 May 4;143(18):1735-1749. doi: 10.1161/CIRCULATIONAHA.120.048740. Epub 2021 Feb 8. PMID 33554616
- [Derived] Sarraju A, Li J, Cannon CP, Chang TI, Agarwal R, Bakris G, Charytan DM, de Zeeuw D, Greene T, Heerspink HJL, Levin A, Neal B, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Perkovic V, Jardine M, Mahaffey KW. Effects of canagliflozin on cardiovascular, renal, and safety outcomes in participants with type 2 diabetes and chronic kidney disease according to history of heart failure: Results from the CREDENCE trial. Am Heart J. 2021 Mar;233:141-148. doi: 10.1016/j.ahj.2020.12.008. Epub 2020 Dec 22. PMID 33358942
- [Derived] Durkin M, Blais J. Linear Projection of Estimated Glomerular Filtration Rate Decline with Canagliflozin and Implications for Dialysis Utilization and Cost in Diabetic Nephropathy. Diabetes Ther. 2021 Feb;12(2):499-508. doi: 10.1007/s13300-020-00953-4. Epub 2020 Dec 18. PMID 33340064
- [Derived] Willis M, Nilsson A, Kellerborg K, Ball P, Roe R, Traina S, Beale R, Newell I. Cost-Effectiveness of Canagliflozin Added to Standard of Care for Treating Diabetic Kidney Disease (DKD) in Patients with Type 2 Diabetes Mellitus (T2DM) in England: Estimates Using the CREDEM-DKD Model. Diabetes Ther. 2021 Jan;12(1):313-328. doi: 10.1007/s13300-020-00968-x. Epub 2020 Dec 2. PMID 33263893
- [Derived] Willis M, Asseburg C, Slee A, Nilsson A, Neslusan C. Development and Internal Validation of a Discrete Event Simulation Model of Diabetic Kidney Disease Using CREDENCE Trial Data. Diabetes Ther. 2020 Nov;11(11):2657-2676. doi: 10.1007/s13300-020-00923-w. Epub 2020 Sep 15. PMID 32930969
- [Derived] Jardine MJ, Zhou Z, Mahaffey KW, Oshima M, Agarwal R, Bakris G, Bajaj HS, Bull S, Cannon CP, Charytan DM, de Zeeuw D, Di Tanna GL, Greene T, Heerspink HJL, Levin A, Neal B, Pollock C, Qiu R, Sun T, Wheeler DC, Zhang H, Zinman B, Rosenthal N, Perkovic V; CREDENCE Study Investigators. Renal, Cardiovascular, and Safety Outcomes of Canagliflozin by Baseline Kidney Function: A Secondary Analysis of the CREDENCE Randomized Trial. J Am Soc Nephrol. 2020 May;31(5):1128-1139. doi: 10.1681/ASN.2019111168. PMID 32354987
- [Derived] Cannon CP, Perkovic V, Agarwal R, Baldassarre J, Bakris G, Charytan DM, de Zeeuw D, Edwards R, Greene T, Heerspink HJL, Jardine MJ, Levin A, Li JW, Neal B, Pollock C, Wheeler DC, Zhang H, Zinman B, Mahaffey KW. Evaluating the Effects of Canagliflozin on Cardiovascular and Renal Events in Patients With Type 2 Diabetes Mellitus and Chronic Kidney Disease According to Baseline HbA1c, Including Those With HbA1c <7%: Results From the CREDENCE Trial. Circulation. 2020 Feb 4;141(5):407-410. doi: 10.1161/CIRCULATIONAHA.119.044359. Epub 2019 Nov 11. No abstract available. PMID 31707795
- [Derived] Mahaffey KW, Jardine MJ, Bompoint S, Cannon CP, Neal B, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Capuano G, de Zeeuw D, Greene T, Levin A, Pollock C, Sun T, Wheeler DC, Yavin Y, Zhang H, Zinman B, Rosenthal N, Brenner BM, Perkovic V. Canagliflozin and Cardiovascular and Renal Outcomes in Type 2 Diabetes Mellitus and Chronic Kidney Disease in Primary and Secondary Cardiovascular Prevention Groups. Circulation. 2019 Aug 27;140(9):739-750. doi: 10.1161/CIRCULATIONAHA.119.042007. Epub 2019 Jul 11. PMID 31291786
- [Derived] Perkovic V, Jardine MJ, Neal B, Bompoint S, Heerspink HJL, Charytan DM, Edwards R, Agarwal R, Bakris G, Bull S, Cannon CP, Capuano G, Chu PL, de Zeeuw D, Greene T, Levin A, Pollock C, Wheeler DC, Yavin Y, Zhang H, Zinman B, Meininger G, Brenner BM, Mahaffey KW; CREDENCE Trial Investigators. Canagliflozin and Renal Outcomes in Type 2 Diabetes and Nephropathy. N Engl J Med. 2019 Jun 13;380(24):2295-2306. doi: 10.1056/NEJMoa1811744. Epub 2019 Apr 14. PMID 30990260
- [Derived] Jardine MJ, Mahaffey KW, Neal B, Agarwal R, Bakris GL, Brenner BM, Bull S, Cannon CP, Charytan DM, de Zeeuw D, Edwards R, Greene T, Heerspink HJL, Levin A, Pollock C, Wheeler DC, Xie J, Zhang H, Zinman B, Desai M, Perkovic V; CREDENCE study investigators. The Canagliflozin and Renal Endpoints in Diabetes with Established Nephropathy Clinical Evaluation (CREDENCE) Study Rationale, Design, and Baseline Characteristics. Am J Nephrol. 2017 Dec 13;46(6):462-472. doi: 10.1159/000484633. Online ahead of print. PMID 29253846

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12900 participants were pre-screened, of those, 8932 were screened. A total of 4401 participants were randomized, with 2199 and 2202 participants assigned to placebo and canagliflozin 100 milligrams (mg), respectively.
Groups:
- Placebo: Participants received matching placebo orally once daily.
- Canagliflozin 100 mg: Participants received canagliflozin 100 milligram (mg) orally once daily.
Period: Overall Study
Arm/Group | Placebo | Canagliflozin 100 mg
Started | 2199 | 2202
Treated | 2197 | 2200
Completed | 2174 | 2187
Not Completed | 25 | 15
Not completed — Closed Site | 1 | 1
Not completed — Withdrawal by Subject | 11 | 5
Not completed — Lost to Follow-up | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Canagliflozin 100 mg | Total
Number analyzed (Participants) | 2199 | 2202 | 4401
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.23) | 62.9 (9.17) | 63 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 732 | 762 | 1494
  Male | 1467 | 1440 | 2907
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 706 | 717 | 1423
  Not Hispanic or Latino | 1457 | 1436 | 2893
  Unknown or Not Reported | 36 | 49 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 452 | 425 | 877
  Black or African American | 112 | 112 | 224
  Hispanic or Latino | 554 | 567 | 1121
  Other | 199 | 189 | 388
  White Non-Hispanic | 882 | 909 | 1791
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 205 | 221 | 426
  AUSTRALIA | 18 | 20 | 38
  BRAZIL | 162 | 152 | 314
  BULGARIA | 13 | 16 | 29
  CANADA | 93 | 79 | 172
  CHILE | 30 | 22 | 52
  CHINA | 63 | 66 | 129
  COLOMBIA | 42 | 52 | 94
  CZECH REPUBLIC | 26 | 31 | 57
  FRANCE | 33 | 28 | 61
  GERMANY | 6 | 5 | 11
  GUATEMALA | 26 | 29 | 55
  HUNGARY | 68 | 67 | 135
  INDIA | 82 | 62 | 144
  ITALY | 39 | 51 | 90
  JAPAN | 53 | 57 | 110
  LITHUANIA | 3 | 4 | 7
  MALAYSIA | 72 | 63 | 135
  MEXICO | 152 | 151 | 303
  NEW ZEALAND | 30 | 31 | 61
  PHILIPPINES | 35 | 36 | 71
  POLAND | 27 | 23 | 50
  ROMANIA | 27 | 32 | 59
  RUSSIAN FEDERATION | 76 | 57 | 133
  SERBIA | 19 | 21 | 40
  SLOVAKIA | 32 | 34 | 66
  SOUTH AFRICA | 34 | 28 | 62
  SOUTH KOREA | 58 | 64 | 122
  SPAIN | 58 | 83 | 141
  TAIWAN | 22 | 15 | 37
  UKRAINE | 173 | 198 | 371
  UNITED ARAB EMIRATES | 0 | 1 | 1
  UNITED KINGDOM | 59 | 59 | 118
  UNITED STATES | 363 | 344 | 707

OUTCOME MEASURES:

1. Primary Outcome: Primary Composite Endpoint of Doubling of Serum Creatinine (DoSC), End-stage Kidney Disease (ESKD), and Renal or Cardiovascular (CV) Death
Description: Primary composite endpoint is the composite of DoSC, ESKD, and renal or CV death. DoSC: from baseline average determination (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). ESKD: as initiation of maintenance dialysis for at least 30 days, or renal transplantation, or an estimated glomerular filtration rate (eGFR) value of less than (<)15 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). Renal death: death in participants who had reached ESKD, died without initiating renal replacement therapy, and no other cause of death was determined via adjudication. Adjudication of these events by Endpoint Adjudication Committee (EAC) was performed in blinded fashion. Event rate estimated based on time to first occurrence of primary composite endpoint are presented.
Time Frame: Up to 4.6 years
Population: The Intent-to-treat (ITT) population consisted of all randomized participants.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 61.24 | 43.21
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p < 0.0001, Cox Proportional Hazard; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.59 to 0.82]

2. Secondary Outcome: Composite Endpoint of CV Death and Hospitalized Heart Failure (HHF)
Description: The composite endpoint included CV death and HHF. CV death included death due to myocardial infarction (MI), stroke, heart failure, sudden death, death during a CV procedure or as a result of procedure-related complications, or death due to other CV causes. For analytic purposes, undetermined causes of death were considered CV deaths. In determining whether a death event was CV in nature, the EAC took into consideration both the proximate and underlying causes. Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of the composite endpoint of CV death and HHF are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 45.44 | 31.47
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0001, Cox proportional hazard; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.57 to 0.83]

3. Secondary Outcome: Major Adverse Cardiac Event (MACE)
Description: The composite endpoint included CV death, non-fatal MI, and non-fatal stroke (that is, 3-point MACE). Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of MACE are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 48.67 | 38.71
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0121, Cox proportional hazard; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.67 to 0.95]

4. Secondary Outcome: Hospitalized Heart Failure (HHF)
Description: Adjudication of these events by the Endpoint Adjudication Committee (EAC) was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of hospitalized heart failure are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 25.33 | 15.65
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0003, Cox proportional hazards; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.47 to 0.80]

5. Secondary Outcome: Renal Composite Endpoint
Description: The renal composite endpoint included composite of DoSC, ESKD and Renal death. DoSC: from the baseline average determination (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). ESKD: initiation of maintenance dialysis for at least 30 days, or renal transplantation, or an eGFR value of <15 mL/min/1.73 m^2 (sustained and confirmed by repeat central laboratory measure after at least 30 days and preferably within 60 days). Renal death: death in participants who have reached ESKD, died without initiating renal replacement therapy, and no other cause of death was determined via adjudication. Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of the renal composite endpoint are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participant.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 40.36 | 26.99
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p < 0.0001, Cox proportional hazards; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.53 to 0.81]

6. Secondary Outcome: Cardiovascular (CV) Death
Description: CV death included death due to MI, stroke, heart failure, sudden death, death during a CV procedure or as a result of procedure-related complications, or death due to other CV causes. For analytic purposes, undetermined causes of death were considered CV deaths. In determining whether a death event was a CV in nature, the EAC took into consideration both the proximate and underlying causes. Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of CV death are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 24.38 | 19.01
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0502, Cox proportional hazards; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.61 to 1.00]

7. Secondary Outcome: All-cause Mortality
Description: Adjudication of these events by Endpoint Adjudication Committee (EAC) was performed in a blinded fashion. Event rate estimated based on time to first occurrence of all-cause mortality are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participants.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 35.00 | 29.04
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0727, Cox proportional hazard; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.02]

8. Secondary Outcome: CV Composite Endpoint
Description: The CV composite endpoint included the CV death, non-fatal MI, non-fatal stroke, hospitalized heart failure, and hospitalized unstable angina. CV death included death due to MI, stroke, heart failure, sudden death, death during a CV procedure or as a result of procedure-related complications, or death due to other CV causes. For analytic purposes, undetermined causes of death were considered CV deaths. In determining whether a death event was a CV in nature, the EAC took into consideration both the proximate and underlying causes. Adjudication of these events by the EAC was performed in a blinded fashion. Event rate estimated based on the time to the first occurrence of the CV composite endpoint are presented.
Time Frame: Up to 4.6 years
Population: The ITT population consisted of all randomized participant.
Measure: Number; unit: Event rate per 1000 participant-years
Arm/Group | Placebo | Canagliflozin 100 mg
Number analyzed (Participants) | 2199 | 2202
Event rate per 1000 participant-years | 66.95 | 49.35
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin 100 mg; Comparison for canagliflozin versus placebo is reported here; Test type: Superiority; p = 0.0001, Cox proportional hazards; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.63 to 0.86]

ADVERSE EVENTS:
Time Frame: Up to 4.6 years
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Canagliflozin 100 mg
All-Cause Mortality (participants affected / at risk) | 193/2197 | 164/2200
Serious Adverse Events (participants affected / at risk) | 806/2197 | 737/2200
Other Adverse Events (participants affected / at risk) | 1447/2197 | 1320/2200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2197) | Canagliflozin 100 mg (N=2200)
Anaemia (Blood and lymphatic system disorders) | 10 | 7
Anaemia Vitamin B12 Deficiency (Blood and lymphatic system disorders) | 0 | 1
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 2 | 2
Hypochromic Anaemia (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Nephrogenic Anaemia (Blood and lymphatic system disorders) | 2 | 1
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Normocytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 8 | 12
Acute Left Ventricular Failure (Cardiac disorders) | 4 | 0
Acute Myocardial Infarction (Cardiac disorders) | 38 | 38
Angina Pectoris (Cardiac disorders) | 14 | 21
Angina Unstable (Cardiac disorders) | 29 | 17
Arrhythmia (Cardiac disorders) | 1 | 2
Arteriosclerosis Coronary Artery (Cardiac disorders) | 3 | 4
Atrial Fibrillation (Cardiac disorders) | 19 | 16
Atrial Flutter (Cardiac disorders) | 2 | 2
Atrioventricular Block (Cardiac disorders) | 2 | 2
Atrioventricular Block Complete (Cardiac disorders) | 2 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 2
Brugada Syndrome (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 7 | 5
Cardiac Asthma (Cardiac disorders) | 1 | 0
Cardiac Disorder (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 50 | 34
Cardiac Failure Acute (Cardiac disorders) | 6 | 6
Cardiac Failure Chronic (Cardiac disorders) | 4 | 2
Cardiac Failure Congestive (Cardiac disorders) | 48 | 24
Cardiac Fibrillation (Cardiac disorders) | 1 | 0
Cardiac Tamponade (Cardiac disorders) | 0 | 1
Cardio-Respiratory Arrest (Cardiac disorders) | 3 | 4
Cardiogenic Shock (Cardiac disorders) | 8 | 2
Cardiomyopathy (Cardiac disorders) | 2 | 0
Cardiorenal Syndrome (Cardiac disorders) | 1 | 1
Chronic Left Ventricular Failure (Cardiac disorders) | 1 | 0
Chronic Right Ventricular Failure (Cardiac disorders) | 1 | 0
Cor Pulmonale (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 23 | 9
Coronary Artery Insufficiency (Cardiac disorders) | 2 | 1
Coronary Artery Occlusion (Cardiac disorders) | 0 | 3
Coronary Artery Stenosis (Cardiac disorders) | 5 | 3
Hypertensive Heart Disease (Cardiac disorders) | 0 | 2
Ischaemic Cardiomyopathy (Cardiac disorders) | 6 | 4
Left Ventricular Failure (Cardiac disorders) | 5 | 3
Mitral Valve Incompetence (Cardiac disorders) | 3 | 1
Myocardial Infarction (Cardiac disorders) | 27 | 22
Myocardial Ischaemia (Cardiac disorders) | 8 | 8
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 2 | 2
Pericardial Haemorrhage (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 1
Pulseless Electrical Activity (Cardiac disorders) | 1 | 1
Right Ventricular Failure (Cardiac disorders) | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 2 | 0
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 2
Ventricular Fibrillation (Cardiac disorders) | 2 | 1
Ventricular Tachycardia (Cardiac disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 2
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 | 1
Thyroid Mass (Endocrine disorders) | 0 | 2
Amaurosis (Eye disorders) | 1 | 0
Angle Closure Glaucoma (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 9 | 8
Cataract Subcapsular (Eye disorders) | 1 | 0
Diabetic Retinopathy (Eye disorders) | 4 | 7
Eye Haemorrhage (Eye disorders) | 3 | 1
Eyelid Ptosis (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 2 | 1
Keratitis (Eye disorders) | 1 | 0
Maculopathy (Eye disorders) | 0 | 2
Neovascular Age-Related Macular Degeneration (Eye disorders) | 1 | 0
Optic Ischaemic Neuropathy (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 2 | 3
Rhegmatogenous Retinal Detachment (Eye disorders) | 1 | 0
Tractional Retinal Detachment (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 1 | 0
Visual Impairment (Eye disorders) | 2 | 1
Vitreous Adhesions (Eye disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 1 | 4
Abdominal Fat Apron (Gastrointestinal disorders) | 0 | 1
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Anal Fistula (Gastrointestinal disorders) | 1 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Chronic Gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diabetic Gastroparesis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Diverticulum (Gastrointestinal disorders) | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 2
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 3 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0
Epulis (Gastrointestinal disorders) | 1 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 1 | 3
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 6 | 4
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 4
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 7
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Large Intestine Polyp (Gastrointestinal disorders) | 2 | 1
Leukoplakia Oral (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Obstructive Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 4
Pancreatitis Acute (Gastrointestinal disorders) | 3 | 3
Peptic Ulcer (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Rectal Polyp (Gastrointestinal disorders) | 0 | 1
Small Intestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 1
Subileus (Gastrointestinal disorders) | 1 | 0
Swollen Tongue (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 2 | 0
Atrophy (General disorders) | 1 | 0
Cardiac Death (General disorders) | 1 | 3
Chest Discomfort (General disorders) | 1 | 1
Chest Pain (General disorders) | 3 | 1
Complication Associated with Device (General disorders) | 0 | 1
Critical Illness (General disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Death (General disorders) | 6 | 7
Drowning (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 0 | 1
General Physical Health Deterioration (General disorders) | 0 | 1
Generalised Oedema (General disorders) | 2 | 2
Incarcerated Hernia (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 1 | 0
Localised Oedema (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 2 | 1
Necrobiosis (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 8
Oedema Peripheral (General disorders) | 4 | 3
Peripheral Swelling (General disorders) | 3 | 1
Pyrexia (General disorders) | 1 | 2
Sudden Cardiac Death (General disorders) | 2 | 2
Sudden Death (General disorders) | 8 | 3
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis Acute (Hepatobiliary disorders) | 0 | 1
Cholangitis Sclerosing (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 5 | 2
Cholecystitis Acute (Hepatobiliary disorders) | 4 | 5
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 3
Cholelithiasis (Hepatobiliary disorders) | 2 | 5
Hepatic Cirrhosis (Hepatobiliary disorders) | 2 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 0 | 1
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 1 | 1
Drug Hypersensitivity (Immune system disorders) | 2 | 0
Abdominal Abscess (Infections and infestations) | 1 | 1
Abdominal Sepsis (Infections and infestations) | 0 | 1
Abdominal Wall Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 3
Acute Hepatitis B (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 3 | 2
Appendicitis Perforated (Infections and infestations) | 3 | 0
Arteriovenous Fistula Site Infection (Infections and infestations) | 2 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 2
Atypical Pneumonia (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial Pyelonephritis (Infections and infestations) | 1 | 0
Bacterial Sepsis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 7 | 5
Bronchitis Viral (Infections and infestations) | 1 | 0
Campylobacter Colitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 26 | 18
Cellulitis Staphylococcal (Infections and infestations) | 1 | 0
Chronic Sinusitis (Infections and infestations) | 2 | 0
Clostridium Difficile Colitis (Infections and infestations) | 1 | 2
Clostridium Difficile Infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 2
Dengue Fever (Infections and infestations) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Diabetic Foot Infection (Infections and infestations) | 4 | 3
Diabetic Gangrene (Infections and infestations) | 2 | 5
Diverticulitis (Infections and infestations) | 2 | 4
Dysentery (Infections and infestations) | 1 | 0
Ear Infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Endophthalmitis (Infections and infestations) | 1 | 0
Enteritis Infectious (Infections and infestations) | 1 | 0
Enterobacter Infection (Infections and infestations) | 0 | 1
Enterocolitis Bacterial (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 5 | 2
Escherichia Sepsis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 15 | 10
Gas Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 19 | 6
Gastroenteritis Bacterial (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Gastrointestinal Bacterial Infection (Infections and infestations) | 1 | 0
Giardiasis (Infections and infestations) | 1 | 0
Graft Infection (Infections and infestations) | 0 | 1
Groin Abscess (Infections and infestations) | 1 | 0
Haemophilus Infection (Infections and infestations) | 0 | 1
Hepatic Echinococciasis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 6 | 5
Infection in An Immunocompromised Host (Infections and infestations) | 1 | 0
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 3
Intervertebral Discitis (Infections and infestations) | 1 | 0
Keratitis Fungal (Infections and infestations) | 2 | 0
Laryngitis (Infections and infestations) | 0 | 1
Liver Abscess (Infections and infestations) | 1 | 0
Localised Infection (Infections and infestations) | 6 | 6
Lower Respiratory Tract Infection (Infections and infestations) | 3 | 2
Lung Infection (Infections and infestations) | 3 | 2
Mediastinitis (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 1 | 0
Meningitis Bacterial (Infections and infestations) | 1 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 2
Onychomycosis (Infections and infestations) | 0 | 1
Opisthorchiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 11 | 11
Osteomyelitis Acute (Infections and infestations) | 0 | 2
Osteomyelitis Chronic (Infections and infestations) | 0 | 1
Perineal Abscess (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 1 | 0
Pharyngeal Abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 86 | 63
Pneumonia Bacterial (Infections and infestations) | 2 | 0
Pneumonia Influenzal (Infections and infestations) | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 3 | 2
Pseudomonas Bronchitis (Infections and infestations) | 1 | 0
Pulmonary Sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 5 | 3
Pyelonephritis Acute (Infections and infestations) | 2 | 4
Pyelonephritis Chronic (Infections and infestations) | 2 | 0
Rectal Abscess (Infections and infestations) | 0 | 1
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 2 | 2
Respiratory Tract Infection Viral (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0
Scrotal Abscess (Infections and infestations) | 1 | 1
Scrub Typhus (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 12 | 11
Septic Shock (Infections and infestations) | 12 | 5
Soft Tissue Infection (Infections and infestations) | 0 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1
Staphylococcal Sepsis (Infections and infestations) | 2 | 2
Streptococcal Infection (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 3
Urinary Tract Infection (Infections and infestations) | 21 | 25
Urinary Tract Infection Fungal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 3 | 3
Viral Infection (Infections and infestations) | 1 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 1 | 6
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 3 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Chest Injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary Artery Reocclusion (Injury, poisoning and procedural complications) | 1 | 0
Coronary Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 | 1
Expired Product Administered (Injury, poisoning and procedural complications) | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 4
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 5
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 2
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Foreign Body in Eye (Injury, poisoning and procedural complications) | 1 | 0
Fracture Displacement (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 5 | 3
Humerus Fracture (Injury, poisoning and procedural complications) | 2 | 4
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle Injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural Intestinal Perforation (Injury, poisoning and procedural complications) | 1 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 2 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 1
Soft Tissue Injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 3 | 3
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 2
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 2
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 0 | 2
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 5 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wound Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Aspiration Bronchial (Investigations) | 0 | 1
Biopsy Kidney (Investigations) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 2
Blood Creatinine Increased (Investigations) | 20 | 7
Blood Glucose Increased (Investigations) | 2 | 1
Blood Osmolarity Decreased (Investigations) | 1 | 0
Blood Urea Increased (Investigations) | 0 | 1
Ejection Fraction Decreased (Investigations) | 1 | 0
Glomerular Filtration Rate Decreased (Investigations) | 1 | 5
Haemoglobin Decreased (Investigations) | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0
Troponin Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 8 | 4
Diabetes Mellitus (Metabolism and nutrition disorders) | 10 | 5
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 12 | 7
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 | 9
Diabetic Ketosis (Metabolism and nutrition disorders) | 1 | 0
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 3 | 1
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 4 | 3
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 1
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 11 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 6 | 2
Metabolic Disorder (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 2
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Displacement (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 5 | 2
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathic Arthropathy (Musculoskeletal and connective tissue disorders) | 3 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis Deformans (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 11 | 10
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 4
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Symphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 2 | 0
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign Neoplasm of Bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Gastric Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large Intestine Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Neoplasm of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Meningioma Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Hodgkin's Lymphoma Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Endometrioid Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Peritoneal Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 8
Prostatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectosigmoid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous Cell Carcinoma of the Vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional Cell Cancer of Renal Pelvis and Ureter Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional Cell Cancer of the Renal Pelvis and Ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amputation Stump Pain (Nervous system disorders) | 1 | 0
Basilar Migraine (Nervous system disorders) | 1 | 1
Brain Injury (Nervous system disorders) | 0 | 1
Brain Oedema (Nervous system disorders) | 0 | 2
Carotid Artery Occlusion (Nervous system disorders) | 1 | 1
Carotid Artery Stenosis (Nervous system disorders) | 8 | 4
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 2
Cauda Equina Syndrome (Nervous system disorders) | 0 | 1
Cerebellar Haemorrhage (Nervous system disorders) | 0 | 1
Cerebellar Infarction (Nervous system disorders) | 1 | 0
Cerebellar Stroke (Nervous system disorders) | 0 | 1
Cerebral Haematoma (Nervous system disorders) | 1 | 1
Cerebral Haemorrhage (Nervous system disorders) | 4 | 1
Cerebral Hypoperfusion (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 7 | 6
Cerebral Ischaemia (Nervous system disorders) | 2 | 2
Cerebrovascular Accident (Nervous system disorders) | 36 | 30
Cervical Radiculopathy (Nervous system disorders) | 1 | 0
Chronic Inflammatory Demyelinating Polyradiculoneuropathy (Nervous system disorders) | 0 | 1
Clonus (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 1 | 2
Depressed Level of Consciousness (Nervous system disorders) | 1 | 0
Diabetic Autonomic Neuropathy (Nervous system disorders) | 0 | 1
Diabetic Hyperosmolar Coma (Nervous system disorders) | 0 | 1
Diabetic Neuropathy (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dural Arteriovenous Fistula (Nervous system disorders) | 1 | 0
Embolic Cerebral Infarction (Nervous system disorders) | 0 | 1
Embolic Stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 0
Facial Paralysis (Nervous system disorders) | 0 | 1
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 1 | 1
Haemorrhagic Stroke (Nervous system disorders) | 4 | 3
Haemorrhagic Transformation Stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0
Hypoglycaemic Encephalopathy (Nervous system disorders) | 1 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 2 | 1
Intracranial Mass (Nervous system disorders) | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 1 | 0
Ischaemic Neuropathy (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 17 | 14
Lacunar Infarction (Nervous system disorders) | 4 | 4
Language Disorder (Nervous system disorders) | 1 | 0
Lumbar Radiculopathy (Nervous system disorders) | 1 | 1
Lumbosacral Radiculopathy (Nervous system disorders) | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 0 | 1
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 | 1
Piriformis Syndrome (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Progressive Supranuclear Palsy (Nervous system disorders) | 1 | 0
Radicular Syndrome (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 0 | 1
Status Epilepticus (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 4
Tension Headache (Nervous system disorders) | 0 | 2
Thalamic Infarction (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 4 | 10
Vascular Encephalopathy (Nervous system disorders) | 2 | 1
Vasculitis Cerebral (Nervous system disorders) | 0 | 1
Vertebral Artery Stenosis (Nervous system disorders) | 1 | 0
Vith Nerve Paralysis (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Retained Products of Conception (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device Malfunction (Product Issues) | 2 | 0
Affective Disorder (Psychiatric disorders) | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 1
Confusional State (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 3 | 1
Disorientation (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0
Substance-Induced Psychotic Disorder (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 50 | 41
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder Cyst (Renal and urinary disorders) | 0 | 1
Calculus Urinary (Renal and urinary disorders) | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 12 | 12
Diabetic Nephropathy (Renal and urinary disorders) | 10 | 12
End Stage Renal Disease (Renal and urinary disorders) | 23 | 16
Glomerulonephritis Chronic (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 4 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 2
Neurogenic Bladder (Renal and urinary disorders) | 0 | 1
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 9 | 5
Renal Impairment (Renal and urinary disorders) | 7 | 10
Renal Injury (Renal and urinary disorders) | 0 | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 1
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urethral Stenosis (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 2
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Acquired Phimosis (Reproductive system and breast disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 4 | 3
Cervix Disorder (Reproductive system and breast disorders) | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0
Genital Swelling (Reproductive system and breast disorders) | 1 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Postmenopausal Haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1
Uterovaginal Prolapse (Reproductive system and breast disorders) | 0 | 1
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Apnoeic Attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dyspnoea at Rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Septum Perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal Cord Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2
Diabetic Foot (Skin and subcutaneous tissue disorders) | 10 | 15
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Idiopathic Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Neuropathic Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 8 | 18
Hospitalisation (Surgical and medical procedures) | 1 | 0
Accelerated Hypertension (Vascular disorders) | 0 | 1
Aortic Dissection (Vascular disorders) | 0 | 1
Aortic Stenosis (Vascular disorders) | 5 | 3
Arterial Disorder (Vascular disorders) | 0 | 1
Arterial Insufficiency (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 3 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 7 | 2
Diabetic Vascular Disorder (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 1 | 0
Embolism Arterial (Vascular disorders) | 2 | 0
Extremity Necrosis (Vascular disorders) | 8 | 9
Haematoma (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 7 | 7
Hypertensive Crisis (Vascular disorders) | 9 | 9
Hypertensive Emergency (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 3 | 4
Intermittent Claudication (Vascular disorders) | 0 | 1
Leriche Syndrome (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 1 | 0
Necrosis Ischaemic (Vascular disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 5 | 2
Peripheral Arterial Occlusive Disease (Vascular disorders) | 11 | 10
Peripheral Artery Occlusion (Vascular disorders) | 0 | 2
Peripheral Ischaemia (Vascular disorders) | 5 | 3
Peripheral Vascular Disorder (Vascular disorders) | 1 | 5
Peripheral Venous Disease (Vascular disorders) | 0 | 1
Post Thrombotic Syndrome (Vascular disorders) | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 0 | 1
Subclavian Artery Stenosis (Vascular disorders) | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 0 | 1
Vascular Occlusion (Vascular disorders) | 0 | 1
Venous Haemorrhage (Vascular disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=2197) | Canagliflozin 100 mg (N=2200)
Anaemia (Blood and lymphatic system disorders) | 136 | 77
Vertigo (Ear and labyrinth disorders) | 50 | 46
Cataract (Eye disorders) | 80 | 58
Diabetic Retinopathy (Eye disorders) | 55 | 65
Constipation (Gastrointestinal disorders) | 82 | 80
Diarrhoea (Gastrointestinal disorders) | 105 | 91
Nausea (Gastrointestinal disorders) | 52 | 54
Vomiting (Gastrointestinal disorders) | 48 | 41
Oedema Peripheral (General disorders) | 199 | 119
Bronchitis (Infections and infestations) | 86 | 83
Gastroenteritis (Infections and infestations) | 51 | 49
Influenza (Infections and infestations) | 88 | 87
Nasopharyngitis (Infections and infestations) | 133 | 130
Onychomycosis (Infections and infestations) | 33 | 45
Pneumonia (Infections and infestations) | 52 | 41
Respiratory Tract Infection (Infections and infestations) | 44 | 19
Upper Respiratory Tract Infection (Infections and infestations) | 117 | 90
Urinary Tract Infection (Infections and infestations) | 185 | 202
Limb Injury (Injury, poisoning and procedural complications) | 45 | 43
Blood Creatinine Increased (Investigations) | 185 | 140
Glomerular Filtration Rate Decreased (Investigations) | 80 | 63
Diabetes Mellitus (Metabolism and nutrition disorders) | 44 | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 74 | 54
Hyperkalaemia (Metabolism and nutrition disorders) | 152 | 129
Hyperuricaemia (Metabolism and nutrition disorders) | 75 | 64
Hypoglycaemia (Metabolism and nutrition disorders) | 227 | 213
Arthralgia (Musculoskeletal and connective tissue disorders) | 83 | 81
Back Pain (Musculoskeletal and connective tissue disorders) | 99 | 94
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 54 | 56
Diabetic Neuropathy (Nervous system disorders) | 69 | 56
Headache (Nervous system disorders) | 65 | 69
Acute Kidney Injury (Renal and urinary disorders) | 51 | 50
End Stage Renal Disease (Renal and urinary disorders) | 52 | 30
Renal Impairment (Renal and urinary disorders) | 61 | 42
Cough (Respiratory, thoracic and mediastinal disorders) | 81 | 80
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 | 35
Skin Ulcer (Skin and subcutaneous tissue disorders) | 70 | 85
Hypertension (Vascular disorders) | 193 | 144
Hypotension (Vascular disorders) | 30 | 57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/91/NCT02065791/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/91/NCT02065791/SAP_001.pdf